CLINICAL TRIAL: NCT01014299
Title: Recruitment Maneuver Increases Oxygenation After Intubation in Hypoxemic ICU Patients: a Randomized Controlled Study
Brief Title: Recruitment Maneuver After Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CHU-0061
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Hypoxemia
Keywords: Intubation; Hypoxemia; Mechanical ventilation; Recruitment maneuver; Acute lung injury; Bacterial translocation; Hypoxemic ICU patients requiring invasive mechanical ventilation
MeSH Terms: conditions — Hypoxia; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Other: Recruitment maneuver — Assigned interventions:
  * No intervention after tracheal intubation (control group)
  * Alveolar recruitment maneuver (RM group) immediately after intubation

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a recruitment maneuver immediately after intubation in hypoxemic patients.

DETAILED DESCRIPTION:
In the intensive care unit (ICU), acute respiratory failure is a common problem. Airway management in critically ill patients usually requires endotracheal intubation after rapid sequence induction. Induction of anesthesia is a well known cause of dramatic changes in respiratory mechanics and gas exchange. Moreover, when the intubation is for respiratory failure, the underlying pathology increases these modifications. The reduction in lung volume results in a deep hypoxemia after intubation. Moreover, mechanical ventilation applied on a collapsed lung increases the risk of ventilator induced lung injury. Recruitment maneuver, which consists of a transient increased in inspiratory pressure, decreases anesthesia-induced lung collapse and hypoxemia. During early acute respiratory failure, RM increases oxygenation and lung volume and may reduce lung oedema. Some authors have suggested the potential benefit of an early RM after induction of anesthesia in operating room. To date, no study has evaluated the short term effect of a recruitment maneuver performed early after intubation in critically ill patients. Therefore, our aim was to ascertain whether RM, performed immediately after intubation, is safe and more effective at reducing hypoxemia than usual management, in hypoxemic patients requiring intubation for invasive ventilation in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* adults who met acute respiratory failure requiring intubation
* adults who met hypoxemia, defined by a PaO2 less than 100 mm Hg under a high FiO2 mask driven by at least 10 L/min oxygen.

Exclusion Criteria:

* encephalopathy
* coma
* cardiac resuscitation
* hyperkaliemia (>5.5 mEq/L)
* acute brain injury and recent thoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Oxygenation (PaO2) measured 5 min after the onset of mechanical ventilation | 5 min after the onset of mechanical ventilation

SECONDARY OUTCOMES:
PaO2 at 30 min after intubation, hemodynamic and microbiologic safety, ICU length of stay, ICU mortality and mechanical ventilation duration. | at 30 min after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Constantin JM, Futier E, Perbet S, Roszyk L, Lautrette A, Gillart T, Guerin R, Jabaudon M, Souweine B, Bazin JE, Sapin V. Plasma neutrophil gelatinase-associated lipocalin is an early marker of acute kidney injury in adult critically ill patients: a prospective study. J Crit Care. 2010 Mar;25(1):176.e1-6. doi: 10.1016/j.jcrc.2009.05.010. Epub 2009 Sep 24. PMID 19781900
- [Derived] Constantin JM, Futier E, Cherprenet AL, Chanques G, Guerin R, Cayot-Constantin S, Jabaudon M, Perbet S, Chartier C, Jung B, Guelon D, Jaber S, Bazin JE. A recruitment maneuver increases oxygenation after intubation of hypoxemic intensive care unit patients: a randomized controlled study. Crit Care. 2010;14(2):R76. doi: 10.1186/cc8989. Epub 2010 Apr 28. PMID 20426859